CLINICAL TRIAL: NCT02765828
Title: Determining the Diagnostic Utility of the Identification of Tongue Involvement in Late-Onset Pompe Disease (LOPD)
Brief Title: Identification of Tongue Involvement in Late-Onset Pompe Disease
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00068729
Record Dates: First submitted 2016-04-22; First posted 2016-05-09 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Myopathy; Neuropathy; Glycogen Storage Disease Type II (Late-onset Pompe Disease)
MeSH Terms: conditions — Muscular Diseases; Glycogen Storage Disease Type II | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Late-Onset Pompe Disease
  Interventions: Other: Observational study
- Acquired/Hereditary Myopathy
  Interventions: Other: Observational study
- Neuropathy
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — The following exams will be done in all cohorts: tongue manual muscle testing (MMT), tongue quantitative muscle testing, tongue ultrasound measurements

SUMMARY:
This purpose of this study is to determine if tongue strength and tongue ultrasound measurements differentiates patients with untreated late-onset Pompe Disease (LOPD) from patients with acquires/hereditary myopathies or neuropathies. It is hypothesized that abnormalities in tongue function and structure in patients with LOPD may be useful in discriminating this condition from others that have similar presentations.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 12 years
* confirmed diagnosis of LOPD and naïve to enzyme-replacement therapy (ERT)
* acquired/hereditary myopathy (e.g., dermatomyositis, polymyositis, inclusion body myositis, limb-girdle muscular dystrophy, distal myopathy, myotonic muscular dystrophy, and other myopathy)
* neuropathy (e.g., peripheral neuropathy, cranial neuropathy, autonomic neuropathy, focal neuropathy)

Exclusion Criteria:

* current use, history within the past two years of use, or eligible but declined use of Lumizyme® enzyme replacement therapy (applicable to LOPD group)
* history of stroke, Parkinson's disease, oculopharyngeal muscular dystrophy, head and neck cancer or radiation treatment to head/neck, or other conditions that commonly affect lingual strength
* inability to follow directions for study participation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prospective participants must have a confirmed diagnosis of late-onset Pompe Disease, acquired/hereditary myopathy, or neuropathy.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Maximal lingual (tongue) strength measured via manual muscle testing (MMT) measured via ordinal scale (see description) | Day 1
  Lingual strength will be rated with a validated 0-4 ordinal scale.
  Score Description
  0 - Normal strength, no weakness.
  1. - Mild weakness. The tongue can be overcome with effort.
  2. - Moderate weakness. Easy to overcome.
  3. - Minimal movement. Unable to protrude to either side.
  4. - No movement detected.
Maximal lingual (tongue) strength measured via quantitative muscle testing (QMT) measured in kilopascals (KPA) | Day 1

SECONDARY OUTCOMES:
Maximal muscle thickness measured with ultrasound assessment in millimeters (mm) | Day 1
  Comprises part of assessment of lingual (tongue) structure via qualitative tongue ultrasound assessment. On-screen calipers will be used to perform measurement.
Echo intensity measured with ultrasound assessment utilizing grayscale analysis | Day 1
  Comprises part of assessment of lingual (tongue) structure via qualitative tongue ultrasound assessment. Echo intensity measurements consist of drawing a box over subcutaneous tissue and muscle areas of interest using the grayscale histogram function. This number will be recorded along with the standard deviation (grayscale analysis).

CONTACTS AND LOCATIONS:
Overall Officials: Harrison Jones, PhD, Principal Investigator — Division of Head and Neck Surgery & Communication Sciences, Duke University Medical Center
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No